CLINICAL TRIAL: NCT01457885
Title: Multi-center Single Arm Phase II Study of Myeloablative Allogeneic Stem Cell Transplantation for Non-remission Acute Myeloblastic Leukemia (AML) Using Clofarabine and Busulfan x 4 (CloBu4) Regimen
Brief Title: Multi-center Study of Myeloablative Allo Stem Cell Transplant for Non-remission AML Using CloBu4 Regimen
Acronym: CloBu4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.038
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloblastic Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CloBu4 regimen (Experimental): After pre-conditioning with CloBu4 (Clofarabine/Busulfan x 4), subjects will receive a peripheral blood stem cell transplant
  Interventions: Drug: Clofarabine/Busulfan x 4; Procedure: Peripheral blood stem cell transplant

INTERVENTIONS:
Drug: Clofarabine/Busulfan x 4 — * Clofarabine IV dose level: 40 mg/m2/day x 5 days
  * Busulfan IV dose level: 3.2 mg/kg daily x 4 days
Procedure: Peripheral blood stem cell transplant — Peripheral blood stem cell transplant, after pre-conditioning drug treatment

SUMMARY:
Although transplant results for AML in complete remission (CR) at the time of transplant have improved, transplant results for non-remission AML have been quite poor. Most multi-center studies have focused on standard risk AML patients and not many studies have been done in this population of patients with non-remission AML. There are a large number of older patients with non-remission AML because the complete remission rate with induction chemotherapy decreases with age. Such older patients do not tolerate conventional full intensity conditioning regimens. Thus, an effective and tolerable conditioning regimen for non-remission AML is a great unmet need for current transplant practice.

From the investigators earlier study, it is suggested that replacing Fludarabine of standard FluBu4 regimen by Clofarabine (a related drug with much more potent anti-leukemia effect) in the transplant conditioning regimen may potentiate the anti-tumor activity of the conditioning regimen without adding significant toxicity, a goal of new conditioning regimen development.

The investigators expect to enroll a total of 75 patients from about fifteen sites. The investigators main objective is to confirm both the safety and efficacy as measured by one-year overall survival, of the CloBu4 combination as full intensity conditioning for non-remission acute myelogenous leukemia.

ELIGIBILITY:
Inclusion Criteria:

Disease Criteria

* AML not in remission at the time of transplant

  * "Not in remission" is defined as "greater than 5.0% bone marrow blasts by aspirate morphology," as determined by a bone marrow aspirate obtained within 2 weeks of study registration.
  * For primary induction failure patients: Patients must have failed at least 2 induction regimens.
  * For patients with relapsed disease: Patients who relapse more than 6 months after preceding remission must fail at least one reinduction regimen to be eligible. For patients in whom the preceding remission is equal to or shorter than 6 months duration, no re-induction regimen is required to qualify for this protocol.
* If the pre-transplant bone marrow aspirate and biopsy are hypoplastic (less than 10% cellularity), and blast percentages cannot be determined, the patient is eligible if the preceding bone marrow met the above criteria.
* Patients with peripheral circulating blasts or patients with extramedullary leukemia are eligible if bone marrow aspirate and biopsy meets the above criteria. Age and Organ Function Criteria
* Age: 2 to 65 years in age.
* Cardiac: LVEF ≥ 40% by MUGA (Multi Gated Acquisition) scan or echocardiogram.
* Pulmonary: FEV1 and FVC capacity) ≥ 40% predicted, DLCO (corrected for hemoglobin) ≥ 40% of predicted.
* Children who are unable to cooperate for pulmonary function tests (PFTs), must have no evidence of dyspnea at rest, no exercise intolerance, and not require supplemental oxygen therapy.
* Renal: Age equal to or older than 12: The estimated creatinine clearance (CrCl) must be equal or greater than 60 mL/min/1.73 m2 as calculated by the Cockcroft-Gault Formula. Age younger than 12: Either estimated or measured CrCl should be greater than 90 ml/min/1.73m2. For estimation, Schwartz formula will be used.
* Hepatic: Serum bilirubin ≤ 1.5 x upper limit of normal (ULN); (AST)/ ALT ≤ 2.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN
* Performance status: Karnofsky ≥ 70%., or Lansky≥70% Consent: All patients must sign informed consent

Exclusion Criteria:

* Active life-threatening cancer requiring treatment other than AML
* Non-compliant to medications.
* No appropriate caregivers identified.
* HIV1 (Human Immunodeficiency Virus-1) or HIV2 positive
* Active life-threatening cancer requiring treatment other than AML
* Uncontrolled medical or psychiatric disorders.
* Uncontrolled infections, defined as positive blood cultures within 72 hours of study entry, or evidence of progressive infection
* Active central nervous system (CNS) leukemia
* Preceding allogeneic HSCT
* Receiving intensive chemotherapy within 21 days of registration.
* Patients with preceding primary myelofibrosis
* Peripheral blasts > 10,000/μL at the time of registration

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shin Mineishi, MD, Study Chair — University of Alabama at Birmingham; John M Magenau, MD, Principal Investigator — University of Michigan, Department of Internal Medicine; Stephen J Forman, MD, Study Chair — City of Hope National Medical Center
Locations (12):
- United States (10):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Washington University at St Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbuilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 Patients were enrolled. Only 74 began treatment. 3 of these patients were pediatric and were left off the subsequent analysis.
Groups:
- CloBu4 Regimen: After pre-conditioning with CloBu4 (Clofarabine/Busulfan x 4), subjects will receive a peripheral blood stem cell transplant
  Clofarabine/Busulfan x 4: - Clofarabine IV, 40 mg/m2/day x 5 days, and Busulfan IV, 3.2 mg/kg daily x 4 days
Period: Overall Study
Arm/Group | CloBu4 Regimen
Started | 74
Completed | 74
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 75 patients were enrolled. Only 74 patients were treated. Of the treated patients, 3 were pediatric and were left off of the analysis. 71 adult patients were analyzed.
Arm/Group | CloBu4 Regimen
Number analyzed (Participants) | 71
Age, Continuous [Median (Full Range); unit: years] | 56 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Non Relapse Mortality (NRM)
Description: Percentage of patients passed without relapse/recurrence at 1 year.
Time Frame: 1 year
Population: 75 patients were enrolled. Only 74 patients were treated. 3 of the 74 patients were pediatric and were therefore left off of analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CloBu4 Regimen
Number analyzed (Participants) | 71
percentage of patients | 21 [12 to 31]

2. Secondary Outcome: The Percentage of Patients Alive at 1 Year
Description: Overall survival was calculated following transplant using a CloBu4 conditioning regimen for patients with non-remission AML
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CloBu4 Regimen
Number analyzed (Participants) | 71
percentage of patients | 32 [22 to 44]

3. Secondary Outcome: Incidence of Relapse
Time Frame: 2 years
Population: 75 patients were enrolled. One patient was not treated. 3 patients were pediatric and therefore left off of this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CloBu4 Regimen
Number analyzed (Participants) | 71
percentage of patients | 55 [42 to 66]

ADVERSE EVENTS:
Description: Adverse events were captured for all patients that were treated with study drug. 75 patients were enrolled and 1 patient was not treated. Only 74 patients were treated.
Arm/Group | CloBu4 Regimen
Serious Adverse Events (participants affected / at risk) | 38/74
Other Adverse Events (participants affected / at risk) | 17/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CloBu4 Regimen (N=74)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 3 (3)
Joint infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 7 (7)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Othe (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CloBu4 Regimen (N=74)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 10 (12)
Nausea (Gastrointestinal disorders) | 12 (15)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (5)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (2)
Allergic reaction (Immune system disorders) | 3 (3)
Catheter related infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 4 (4)
Infections and infestations - Other (Infections and infestations) | 3 (9)
Lung infection (Infections and infestations) | 2 (2)
Nail infection (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 3 (3)
Soft tissue infection (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (2)
Investigations - Other, specify (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (3)
Platelet count decreased (Investigations) | 2 (8)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (9)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 2 (2)
Vascular disorders - Other (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes